CLINICAL TRIAL: NCT04710745
Title: Atrial Fibrillation in Relationship to Plasma Biomarkers
Acronym: AFISBIO II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Premedix Academy (Other)
Responsible Party: Sponsor
Other Study IDs: 0012020
Record Dates: First submitted 2021-01-10; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Plasmatic Biomarkers; ECG Monitoring
MeSH Terms: conditions — Atrial Fibrillation | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients in sinus rhythm without history of AF, with high risk for ischemic stroke and AF. CHA2DS2-VASc score > 2 (for females > 3) and with more than 3 specific criteria for inclusion.
  Interventions: Diagnostic Test: Peripheral blood samples for routine analysis including NT-proBNP and plasmatic biomarkers.; Diagnostic Test: Echocardiography; Diagnostic Test: ECG Holter monitor; Diagnostic Test: Standardized Mini-Mental Status Exam (SMMSE)

INTERVENTIONS:
Diagnostic Test: Peripheral blood samples for routine analysis including NT-proBNP and plasmatic biomarkers. — Sampling of peripheral venous blood for analysis of plasma concentration of plasmatic markers (Apelin, microRNA, FGF-23, IGF-1, IGFBP-1) and routine analysis (laboratory parameters: NT-proBNP, D-dimer, Creatinine Clearance, CRP, Hs-troponin).
Diagnostic Test: Echocardiography — ECHO parameters:
  * E/e´
  * Mean e' septal and lateral wall
  * LA volume (Biplane Area-Length Method)
  * Left atrial volume index
  * Diameter of left atrium in PLAX
  * Severe aortic stenosis
  * Severe mitral regurgitation
  * Severe tricuspid regurgitation
  * Left ventricular end-diastolic diameter
  * Interventricular septum
  * Posterior wall
  * LV Mass
  * Left ventricular mass index
Diagnostic Test: ECG Holter monitor — Patient receives an ECG Holter for a 7-day monitoring.
Diagnostic Test: Standardized Mini-Mental Status Exam (SMMSE) — A screening test for evaluating cognitive performance of patients done in the clinician's office.

SUMMARY:
The general objective of this study is to:

A. To identify novel plasmatic biomarkers associated with prevalent/incident atrial fibrillation in patients with high risk for AF and stroke.

B. To assess predictive ability of novel plasmatic biomarkers (especially apelin and miRNAs) on prevalent/incident atrial fibrillation in patients with high risk for AF and stroke.

C. To validate predictive models from previous studies based on comorbidities, age, sex, BMI, NT-proBNP, FGF-23, IGF-1 and IGFBP-1 on prevalent/incident AF in patients with high risk for AF and stroke.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained arrhythmia, associated with an increased risk of stroke, heart failure, and mortality. Despite the high prevalence, AF may be asymptomatic and consequently unrecognized. Detection of asymptomatic AF is challenging as only a minority of the patients is diagnosed during standard examinations with a 12 - lead ECG or a 24h ECG Holter monitoring. Furthermore, prolonged ECG monitoring is costly and can be inconvenient for the patients. Documented AF causes 15% of ischemic strokes. However, approximately 25% of ischemic strokes is of an unknown etiology. It is believed that undetected asymptomatic AF is responsible for some of these strokes.

Plasmatic biomarkers might be of importance in the early diagnosis of AF. Several plasmatic biomarkers have been studied in order to find an association with AF. Cardiac biomarkers such as natriuretic peptides and high-sensitivity troponins are increased in patients with AF. A novel biomarker that is depending on left atrial stretching and ionotropic effects is apelin. In our previous research we discovered that apelin is associated with AF, negatively correlates with AF burden, but only in patients without reduced LVEF. Similarly, parameters reflecting thrombogenesis, such as Fibrinogen and fibrin D-dimer were also found to be associated with the arrhythmia. Other protein biomarkers have been studied in relation to AF incidence. Insulin-like growth factor-binding protein 1 (IGFBP-1) and Insulin-like growth factor 1 (IGF-1) have shown an association with higher risk of incident AF. Previous research also indicated Fibroblast growth factor 23 (FGF-23) to be associated with AF.

However, biomarkers, such as the inflammatory markers high-sensitivity CRP have shown conflicting results.

Finally, in the last years, circulating microRNAs emerged as a promising biomarker of AF, having important function in suppression of messenger RNA responsible for electric and structural remodeling of the left atria.

In our previous case-matched study we discovered that selected miRNAs were associated with paroxysmal AF.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria:

* AGE > 50 years
* No history of supraventricular arrhythmia
* Sinus rhythm at inclusion
* CHADSVASc score > 2 in men (> 3 in female)
* More than 3 specific criteria for inclusion
* Written informed consent is obtained before any study-related assessment is performed

Specific inclusion criteria:

* Age > 65
* Age > 75
* BMI > 30
* Heart failure with preserved LVEF (according to ESC GL for HF)
* Ischemic stroke
* Left atrial diameter > 45mm
* Chronic obstructive pulmonary disease
* Arterial hypertension
* PR interval > 200ms
* History of MI or (objective evidence of) chronic coronary syndrome
* Peripheral artery disease
* Thyroid disease

Exclusion Criteria:

* History of any supraventricular or ventricular arrhythmia (excluding premature contractions and 1st degree AV block)
* Therapy with anticoagulants at the time of inclusion
* Acute coronary syndrome less than 1 month prior to inclusion
* History of cardiac surgery
* Diabetes mellitus type 2
* Reduced LVEF (<50%)
* Acute or decompensated heart failure at the time of inclusion
* Cardiomyopathy
* Systemic inflammatory disease or acute inflammatory disease
* Active malignancy
* Alcoholism (≥ 8 drinks/week)
* Renal Disease (Dialysis/ transplant/ CrCl < 1ml/s)
* Liver disease (cirrhosis/ transaminase > 3x ULT/ bilirubin > 2x ULT)
* Severe or moderate mitral stenosis
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Slovak hospitals and outpatient clinics in sinus rhythm without history of AF, with high risk for ischemic stroke and AF. CHA2DS2-VASc score > 2 (for females > 3) and with more than 3 specific criteria for inclusion.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of AF | Within 14 days from Inclusion.
  AF duration > 30s on surface ECG
Incidence of AF | Within 14 days from Inclusion.
  AF duration > 30s on surface ECG

SECONDARY OUTCOMES:
Cardiovascular (CV) death | Day 175-205 from inclusion (Follow-up 3) - Day 1080-1110 from inclusion (Follow-up 6)
  Event occurred or did not occur (Yes/No).
All cause death | Day 175-205 from inclusion (Follow-up 3) - Day 1080-1110 from inclusion (Follow-up 6)
  Event occurred or did not occur (Yes/No).
CV death + nonfatal stroke + nonfatal myocardial infarction | Day 175-205 from inclusion (Follow-up 3) - Day 1080-1110 from inclusion (Follow-up 6)
  Event occurred or did not occur (Yes/No).
Ischemic stroke | Day 175-205 from inclusion (Follow-up 3) - Day 1080-1110 from inclusion (Follow-up 6)
  Event occurred or did not occur (Yes/No).
Cognitive decline assessed by Mini-Mental State Examination | Day 350-380 from inclusion (Follow-up 4) - Day 1080-1110 from inclusion (Follow-up 6)
  Impairment observed and recorded or not observed and not recorded (Yes/No).
Heart failure | Day 175-205 from inclusion (Follow-up 3) - Day 1080-1110 from inclusion (Follow-up 6)
  Event occurred or did not occur (Yes/No). If Yes, HF classification to be indicated based on LVEF:
  i. with preserved LVEF (HFpEF) ii. with mid-range LVEF (HFmrEF) iii. with reduced LVEF (HFrEF)
Hospitalization due to CV cause | Day 175-205 from inclusion (Follow-up 3) - Day 1080-1110 from inclusion (Follow-up 6)
  Event occurred or did not occur (Yes/No).
Acute coronary syndrome | Day 175-205 from inclusion (Follow-up 3) - Day 1080-1110 from inclusion (Follow-up 6)
  Event occurred or did not occur (Yes/No). If Yes, type of ACS to be indicated:
  i. Unstable angina ii. NSTEMI iii. STEMI

CONTACTS AND LOCATIONS:
Locations (6):
- Slovakia (6):
  - University Hospital Bratislava - Old Town Hospital, Bratislava
  - University Hospital Bratislava - Hospital Ruzinov, Bratislava
  - University Hospital Bratislava - Hospital of the Academician Ladislav Dérer, Bratislava
  - National Institute for Cardiovascular Diseases, Bratislava
  - Hospital Malacky, Malacky
  - Faculty Hospital Nitra, Nitra

IPD SHARING:
Plan to Share IPD: No